CLINICAL TRIAL: NCT02024620
Title: Evaluation of Mood Coach in the Treatment of Major Depressive Disorder
Brief Title: Mobile Apps for the Treatment of Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The mobile phone app upon which the study was based was not available.
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: National Center for PTSD (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 529128
Record Dates: First submitted 2013-12-04; First posted 2013-12-31 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; technology; psychotherapy; behavioral activation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral activation plus mobile app (Experimental): Standard behavioral activation protocol with the addition of the Mood Coach mobile app to replace the paper and pencil forms used in the standard protocol.
  Interventions: Behavioral: Behavioral activation plus mobile app
- Standard behavioral activation (Active Comparator): Standard behavioral activation protocol using paper and pencil forms for treatment delivery and homework completion.
  Interventions: Behavioral: Standard behavioral activation

INTERVENTIONS:
Behavioral: Behavioral activation plus mobile app
  Arms: Behavioral activation plus mobile app
Behavioral: Standard behavioral activation
  Arms: Standard behavioral activation

SUMMARY:
Smartphone applications (apps) may be well-suited as a low cost adjunctive tool for increasing the adherence of individuals to psychotherapy treatments which may subsequently increase symptom reduction and improve clinical outcomes. Apps offer the opportunity for real-time tracking of behavior and have the ability to provide prompt feedback and reminders in a convenient, readily available technology. The immediacy and convenience of apps may be responsible for the observed improvements in adherence on the part of the patients relative to traditional paper-and-pencil tracking and practice of skills taught in psychotherapy. These features are relevant to behavioral activation (BA) protocols, the effects of which are often attenuated by failure to adhere to regular practice and tracking of behavior. The Mood Coach app is a BA protocol developed to provide a convenient means of planning and tracking activity, and monitoring mood responses to scheduled increases in activity. This project evaluates the utility of this app as an adjunct to standard BA treatment. The investigators predict that participants assigned to the BA+app condition will demonstrate greater adherence to the BA treatment compared to the standard BA condition. The investigators also predict that the participants in the BA+app condition will report greater satisfaction with the app compared to the standard BA protocol that utilizes paper and pencil materials.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 18 and older
* Speak and understand English
* Meet criteria for major depressive disorder
* Willing to participate in psychotherapy for depression

Exclusion Criteria:

* Current psychotic disorder diagnosis
* Current bipolar disorder
* Diagnosed with a substance use disorder that is not currently being addressed by a non-study provider
* Patients receiving a concurrent evidence-based psychotherapy for depression or PTSD

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Activation for Depression Scale-Short Form | Week 1, Week 4, Week 8
  Measures symptoms of depression consistent with a behavioral deficits model in a brief format.

SECONDARY OUTCOMES:
Change in Depression Anxiety Stress Scales-21 | Week 1, Week 4, Week 8
  Assesses symptoms of depression, anxiety, and stress in a brief format.

OTHER OUTCOMES:
Homework Compliance Rating Scale | Week 4, Week 8
  Assesses the amount of effort put into the weekly behavioral activation homework. Completed by the participant and the study clinician.
Treatment Evaluation Inventory-Short Form | Week 4, Week 8
  Assesses the degree to which the treatment provided in the project is deemed acceptable by the participant. The measure used in the present project is modified from the original to better assess the treatment procedures in an adult population.
Perceptions of Computerized Therapy Questionnaire-Patient Version | Week 1, Week 8
  Measures participants' opinion of computerized and computer-assisted psychotherapy.
Mini-International Neuropsychiatric Interview | Week 1, Week 8
  Clinician-administered brief diagnostic interview for psychiatric diagnoses. The selected sections for this project include the major depressive disorder, dysthymic disorder, bi-polar disorder, panic disorder, obsessive-compulsive disorder, generalized anxiety, disorder, social anxiety disorder, post-traumatic stress disorder, and substance use disorder sections.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Brady, Ph.D., Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- Central Arkansas Veterans Healthcare System, North Little Rock, Arkansas, United States

REFERENCES:
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Newman MG, Szkodny LE, Llera SJ, Przeworski A. A review of technology-assisted self-help and minimal contact therapies for anxiety and depression: is human contact necessary for therapeutic efficacy? Clin Psychol Rev. 2011 Feb;31(1):89-103. doi: 10.1016/j.cpr.2010.09.008. Epub 2010 Oct 14. PMID 21130939